CLINICAL TRIAL: NCT00023569
Title: Cortical Motor Reorganization in Chronic Stroke Following EMG Triggered NMES Therapy
Brief Title: Electrical Stimulation to Improve Hand Function in Patients With Chronic Stroke
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010248; 01-N-0248
Record Dates: First submitted 2001-09-08; First posted 2001-09-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-09

CONDITIONS: Cerebrovascular Accident
Keywords: TMS; Conjoint Movement; Chronic Hemiplegia; Brain Plasticity; Electrical Stimulation; Stroke; CVA
MeSH Terms: conditions — Stroke

SUMMARY:
This study will determine whether an electric shock to the forearm can improve hand function in patients with chronic stroke and, if so, whether the improvement is related to brain reorganization. Some studies indicate that electromyography-triggered neuromuscular electrical stimulation (EMG-triggered NMES) on the forearm improves wrist motor function in patients with chronic stroke. The shock is delivered to the wrist extensor muscle of the forearm, causing greater hand movement than the patient can make on his or her own. The study will determine if the electric shock is more effective given after the patient initiates the hand movement (EMG-triggered NMES) than at times unrelated to patient effort (NMES alone).

Stroke patients with muscle weakness on one side of the body may be eligible for this study. The stroke must have occurred at least 12 months before the patient enters the study. Candidates will have a medical history and physical and neurological examinations.

Participants will be divided randomly into two groups: EMG-triggered NMES, and NMES alone. For EMG-triggered NMES, two electrodes from the NMES machine and two EMG electrodes are placed on the wrist extensor muscle of the forearm. The patient relaxes the hand, then contracts the wrist extensor muscle to produce movement. This movement triggers the NMES to deliver enough electrical stimulation to produce maximum wrist extension. For NMES alone, only the two NMES electrodes are placed on the forearm. The patient relaxes the hand and stimulation is applied at an intensity to produce full wrist extension without any patient effort.

At the first clinic visit, baseline hand function is measured with the following tests:

* Wrist extension - wrist extension is measured with a digital instrument called an accelerometer
* Pinch power - grip strength between thumb and index finger is measured with a digital pinch analyzer
* Jebsen-Taylor hand function - function is evaluated through activities such as moving a can and lifting a pin
* H reflex - (Note: I could not find a description of this test or its purpose in the consent or the protocol)

In addition, transcranial magnetic stimulation (TMS) is done to examine brain activity. For this test, an insulated wire coil is placed on the patient's scalp. A brief electrical current passes through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the outer part of the brain. The stimulation may cause muscle, hand or arm twitching, or may affect movement or reflexes. During the stimulation, electrical activity of muscles are recorded with a computer or other recording device, using electrodes attached to the skin with tape.

Participants will be instructed in how to use the NMES machine at the first visit. They will be required to practice with the machine at home 30 minutes twice a day every day for 4 weeks, for a total of about 56 sessions. Follow-up evaluations of hand function will be done one day after the first NMES or EGM-triggered NMES task, then after 2 weeks and after 4 weeks of performing the exercise. These evaluations include the tests described above for baseline measurements, plus TMS.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of a newly developed electrical technique, electromyography (EMG) triggered neuromuscular electrical stimulation NMES) known as EMG-Stim., on brain reorganization. Clinically EMG-Stim. is thought to improve a chronic hemiparetic hand [1-3], but its underlying mechanism is poorly understood. We plan to determine: (1) if EMG-Stim. on a chronic hemiparetic hand as a result of stroke enhances improved hand motor function; and (2) whether any clinical improvement is related to brain reorganization.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects with residual arm function who have had a single cortical monohemispheric stroke (documented by CT or MRI) at least 12 months before, with normal visual acuity (with or without glasses).

EXCLUSION CRITERIA

Subjects with more than one stroke.

Subjects with proprioceptive deficits.

Subjects with cerebellar lesion.

Subjects unable to extend metacarpophalangeal (MP) joints at least 10 degrees.

Subjects unable to extend the wrist 10 degrees.

Subjects with cognitive impairment which might interfere with the understanding of instructions for motor testing (defined as equivalent to a mini-mental state exam score of 20 or less).

Subjects with severe depression, poor motivational capacity, or severe language disturbance.

Subjects with severe uncontrolled medical problems (e.g. cardiovascular disease, active joint deformity of arthritic origin, uncontrolled epilepsy).

Subjects with heart pacemakers.

Subjects with contractures in the hand.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2001-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kraft GH, Fitts SS, Hammond MC. Techniques to improve function of the arm and hand in chronic hemiplegia. Arch Phys Med Rehabil. 1992 Mar;73(3):220-7. PMID 1543423
- [Background] Fields RW. Electromyographically triggered electric muscle stimulation for chronic hemiplegia. Arch Phys Med Rehabil. 1987 Jul;68(7):407-14. PMID 3496865
- [Background] Cauraugh J, Light K, Kim S, Thigpen M, Behrman A. Chronic motor dysfunction after stroke: recovering wrist and finger extension by electromyography-triggered neuromuscular stimulation. Stroke. 2000 Jun;31(6):1360-4. doi: 10.1161/01.str.31.6.1360. PMID 10835457